CLINICAL TRIAL: NCT01549665
Title: Umbilical Cord Blood-derived Mesenchymal Stem Cells for the Treatment of Steroid-refractory Acute or Chronic Graft-versus-host-disease
Acronym: GVHD-MSC
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Collaborators: Medipost Co Ltd. (Industry)
Responsible Party: Principal Investigator, Hong Hoe Koo, MD, PhD, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MP-CR-008
Record Dates: First submitted 2012-02-23; First posted 2012-03-09 (Estimated); Last update posted 2012-03-16 (Estimated); Status verified 2012-03

CONDITIONS: Graft-Versus-Host Disease; GVHD; Allogeneic Hematopoietic Transplant; Disorder Related to Transplantation
Keywords: Graft-Versus-Host Disease; GVHD; Hematopoietic Stem Cell Transplantation; Stem Cell Transplantation; Allogeneic hematopoietic transplant; Mesenchymal Stem Cells; Unrelated Donors; Cord Blood Stem Cell Transplantation
MeSH Terms: conditions — Graft vs Host Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: Human umbilical cord blood-derived mesenchymal stem cells — 1st infusion(1x1,000,000 hMSC/kg)IV, 2nd infusion(2x1,000,000 hMSC/kg)IV and 3rd infusion(3x1,000,000 hMSC/kg)IV if no complete response at 28 days.
  Other Names: PROMOSTEM®

SUMMARY:
Graft-versus-host-disease (GVHD) is a major complication following allogeneic hematopoietic stem cell transplantation (allo-HSCT) which may cause acute life-threatening morbidity or chronic disabilities. Although corticosteroid, the primary agent to treat GVHD, may be effective for some patients, outcomes of those who are refractory to corticosteroid are dismal. Secondary agents can be used for steroid-refractory cases; however, their efficacy is variable and usually limited. The quality of life issue of chronic GVHD is especially important for pediatric survivors who have longer life expectancy than adults. Many in-vitro and in-vivo data support immunoregulatory properties of mesenchymal stem cells(MSCs)and possibilities of treating diseases caused by immune dysregulation such as GVHD. Recent data revealed that bone marrow-derived MSCs were very useful to treat steroid-refractory acute GVHD, which led to improved overall survival compared with controls. More recently, a number of reports suggest MSCs may also be useful in treating chronic GVHD as well as acute GVHD. It has been also reported that third party MSCs are also useful as well as those from autologous or HLA-matched donors. The investigator recently demonstrated that MSCs obtained from umbilical cord blood (UCB) have similar immunosuppressive properties as bone marrow-MSCs. UCB-MSCs can be obtained without doing any harm to donors that it may be more appropriate source of MSCs than bone marrow for off-the-shelf use. However, little is known about the safety and efficacy of UCB-MSCs in treating GVHD. Therefore, the investigator designed this study to evaluate the safety and efficacy of UCB-MSCs in treating pediatric patients with steroid-refractory acute or chronic GVHD.

ELIGIBILITY:
Inclusion Criteria:

* Steroid-refractory acute or chronic graft-versus-host-disease
* Acquisition of consent form
* 0-30 years of age

Exclusion Criteria:

* Withdrawal from the study
* Progression of underlying hematologic diseases
* Severe adverse effects related to the investigational drug

Ages: 1 Day to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2012-01; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Safety of UCB-MSC in SR-GVHD | 180 days
  * Vital sign
  * Physical examination
  * ECOG performance status
  * Mixed Lymphocyte Reaction(MLR)
  * Adverse effects related to infusion

SECONDARY OUTCOMES:
Complete, Partial Response Rate at 28 and 180 Days in participants with SR-GVHD treated with UCB-MSC | 180 Days
  * Complete Response(CR) rate(%) = (Number of CR/Number of Participants)x100
  * Partial Response(PR)rate(%) = (Number of PR/Number of Participants)x100

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Pediatrics, Samsung Medical Center, Seoul, South Korea